CLINICAL TRIAL: NCT06628362
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Phase 2 Study to Evaluate the Efficacy, Safety, and Tolerability of Once-Weekly CT-388 Administered Subcutaneously for 48 Weeks to Participants Who Are Overweight or Obese With Type 2 Diabetes Mellitus
Brief Title: A Study of CT-388 in Participants Who Are Overweight or Obese With Type 2 Diabetes Mellitus
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Carmot Therapeutics, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-388-104; XC45544 (Other: Roche Protocol Number)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Overweight or Obese; Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 2: CT-388 Dose Level 1 (Low) (Experimental)
  Interventions: Drug: CT-388
- Arm 3: CT-388 Dose Level 2 (Experimental)
  Interventions: Drug: CT-388
- Arm 4: CT-388 Dose Level 3 (Experimental)
  Interventions: Drug: CT-388
- Arm 5: CT-388 Dose Level 4 (High) (Experimental)
  Interventions: Drug: CT-388

INTERVENTIONS:
Drug: Placebo — Placebo will be volume-matched and administered subcutaneously (SC) once weekly.
  Arms: Arm 1: Placebo
Drug: CT-388 — CT-388 will be administered subcutaneously (SC) once weekly at the randomized dosing regimen.
  Other Names: RO7795068; RG6640
  Arms: Arm 2: CT-388 Dose Level 1 (Low); Arm 3: CT-388 Dose Level 2; Arm 4: CT-388 Dose Level 3; Arm 5: CT-388 Dose Level 4 (High)

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel group dose-finding study to evaluate the efficacy and safety of CT-388 at low, middle, and high doses in participants who are overweight or obese with Type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Body mass index (BMI) ≥25.0 kg/m^2
* Have a diagnosis of Type 2 Diabetes Mellitus (T2DM) according to the World Health Organization classification or other locally applicable standards
* Have an HbA1c ≥7% and ≤10.5%
* Management of T2DM with diet and exercise alone, metformin, or a sodium-glucose cotransporter-2 (SGLT-2) inhibitor, as monotherapy or in combination, per approved local label
* At least one self-reported unsuccessful diet/exercise effort to lose body weight

Exclusion Criteria:

* Have Type 1 Diabetes Mellitus (T1DM), history of ketosis or hyperosmolar state/coma, or any other types of diabetes except T2DM
* Have had 1 or more episodes of Level 3 hypoglycemia or have had hypoglycemia unawareness within 3 months prior to screening
* Have history or presence of proliferative diabetic retinopathy, diabetic macular edema, or non-proliferative diabetic retinopathy that requires acute treatment
* Have evidence of clinically significant autonomic neuropathy (symptoms may include resting tachycardia, orthostatic hypotension, or diabetic diarrhea)
* Had treatment with any oral antihyperglycemic medications, with the exception of metformin or SGLT-2 inhibitors, within 3 months prior to screening or planned concurrent treatment with these medications during the study
* Had treatment with injectable antihyperglycemic medication, with the exception of short-term insulin, within 6 months prior to screening or planned concurrent treatment with these medications during the study
* Self-reported body weight change of >5 kg within 3 months before screening
* Any unbalanced/extreme diets, such as very low calorie, low carbohydrate, very high protein, ketogenic, or intermittent diets, within 3 months of the screening visit, or plan to be on such diets during the study
* Current or recent use of any treatment that promotes weight loss or glucose metabolism
* Current or recent use of treatment that may cause weight gain
* Prior or planned surgical treatment or procedure for obesity, except for liposuction or abdominoplasty if performed >1 year prior to screening. Participants with a history of devices, such as LAP-BAND® or intragastric balloon, are permitted, if devices were removed >1 year prior to screening.
* History of clinically significant or active gastric emptying abnormality (e.g., severe gastroparesis or gastric outlet obstruction, intestinal obstruction), or chronic use of medications that directly affect GI motility
* History of chronic pancreatitis or acute pancreatitis or have signs and symptoms of acute pancreatitis at screening
* Have obesity induced by other endocrinologic disorders (e.g., Cushing syndrome) or diagnosed monogenetic or syndromic forms of obesity
* History or diagnosis of significant active or unstable major depressive disorder or any history/diagnosis of other severe psychiatric conditions (e.g., schizophrenia; bipolar disorder; other serious mood disorder or anxiety disorder, or hyperactivity disorder) within the last year before screening
* History of any hematologic conditions that may interfere with HbA1c measurement (e.g., hemolytic anemias, sickle cell disease, other hemoglobinopathies)
* Family or personal history of medullary thyroid carcinoma
* Women who are pregnant, breastfeeding, or intend to become pregnant, or are of childbearing potential and not using a highly effective contraceptive method as required per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Body Weight from Baseline to Week 36 | Baseline to Week 36
Change in Glycated Hemoglobin (HbA1c) from Baseline to Week 36 | Baseline to Week 36

SECONDARY OUTCOMES:
Percent Change in Body Weight from Baseline to Week 48 | Baseline to Week 48
Change in HbA1c from Baseline to Week 48 | Baseline to Week 48
Percentage of Participants with HbA1c <7.0% at Weeks 36 and 48 | Weeks 36 and 48
Percentage of Participants with Body Weight Reduction ≥5%, ≥10%, ≥15%, ≥20%, and ≥25% from Baseline to Week 36 | Baseline and Week 36
Percentage of Participants with Body Weight Reduction ≥5%, ≥10%, ≥15%, ≥20%, and ≥25% from Baseline to Week 48 | Baseline and Week 48
Percent Change in Body Weight from Baseline to Week 28 | Baseline and Week 28
Absolute Change in Body Weight (kg) from Baseline to Weeks 36 and 48 | Baseline to Weeks 36 and 48
Percent Change in Body Weight from Baseline to Weeks 16, 28, 36, and 48 by Obesity Class | Baseline to Weeks 16, 28, 36, and 48
Change in HbA1c from Baseline to Weeks 16 and 28 | Baseline to Weeks 16 and 28
Change in HbA1c from Baseline to Weeks 16, 28, 36, and 48 by Obesity Class | Baseline to Weeks 16, 28, 36, and 48
Percentage of Participants with HbA1c ≤6.5% at Weeks 16, 28, 36, and 48 | Weeks 16, 28, 36, and 48
Percentage of Participants with HbA1c <5.7% at Weeks 16, 28, 36, and 48 | Weeks 16, 28, 36, and 48
Change in 7-point Self-Monitored Blood Glucose (SMBG) Profile at Weeks 16, 28, 36, and 48 | Weeks 16, 28, 36, and 48
Percentage of Participants who Achieve HbA1c ≤6.5% and ≥10.0% Weight Reduction at Weeks 16, 28, 36, and 48 | Baseline, Weeks 16, 28, 36, and 48
Percentage of Participants who Achieve HbA1c <7.0% and ≥5.0% Weight Reduction at Weeks 16, 28, 36, and 48 | Baseline, Weeks 16, 28, 36, and 48
Change in Body Mass Index (BMI) from Baseline to Weeks 36 and 48 | Baseline, Weeks 36 and 48
Change in Waist Circumference from Baseline to Weeks 36 and 48 | Baseline, Weeks 36 and 48
Change in Hip Circumference from Baseline to Weeks 36 and 48 | Baseline, Weeks 36 and 48
Change in Waist-to-Hip Ratio from Baseline to Weeks 36 and 48 | Baseline, Weeks 36 and 48
Change in Waist-to-Height Ratio from Baseline to Weeks 36 and 48 | Baseline, Weeks 36 and 48
Change in Fasting Plasma Glucose from Baseline to Weeks 16, 28, 36, and 48 | Baseline to Weeks 16, 28, 36, and 48
Change in Fasting Insulin from Baseline to Weeks 16, 28, 36, and 48 | Baseline to Weeks 16, 28, 36, and 48
Change in Fasting C-peptide from Baseline to Weeks 16, 28, 36, and 48 | Baseline to Weeks 16, 28, 36, and 48
Change in Fasting Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) from Baseline to Weeks 16, 28, 36, and 48 | Baseline to Weeks 16, 28, 36, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Carmot Therapeutics, Inc., a Member of the Roche Group
Locations (70):
- United States (52):
  - Central Alabama Research, Birmingham, Alabama
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Lakeview Clinical Research, LLC, Guntersville, Alabama
  - Yuma Clinical Trials, Yuma, Arizona
  - AMCR Institute, Escondido, California
  - Ark Clinical-Fountain Valley, Fountain Valley, California
  - Orange Country Research Center, Lake Forest, California
  - Ark Clinical Research, Long Beach, California
  - Catalina Research Institute, LLC, Montclair, California
  - Asclepes Research Centers, Sherman Oaks, California
  - Encompass Clinical Research, Spring Valley, California
  - Flourish Research - Boca Raton, Boca Raton, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - K2 Medical Research, LLC - Maitland, Maitland, Florida
  - K2 Medical Research, LLC - Orlando, Maitland, Florida
  - Flourish Research Acquisition, LLC, Miami, Florida
  - K2 Medical Research, LLC - South Orlando, Orlando, Florida
  - Aging Well Associates, St. Petersburg, Florida
  - K2 Medical Research Tampa, Tampa, Florida
  - K2 Summit Research, The Villages, Florida
  - Privia Medical Group Georgia, LLC, Fayetteville, Georgia
  - Privia Medical Group Georgia - Thomasville, Thomasville, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Duly Health and Care, Lombard, Illinois
  - McFarland Clinic, Ames, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - NOLA Cares, LLC, Metairie, Louisiana
  - Flourish Research Acquisition, LLC dba Flourish Bowie, Bowie, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - NECCR PrimaCare Research LLC, Fall River, Massachusetts
  - Olive Branch Family Medical Center; Family Medicine, Olive Branch, Mississippi
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Ellipsis Research Group, Brooklyn, New York
  - Accellacare of Cary, Cary, North Carolina
  - Accellacare - Hickory, Hickory, North Carolina
  - Accellacare of Rocky Mount, Rocky Mount, North Carolina
  - Accellacare of Piedmont Healthcare, Statesville, North Carolina
  - Accellacare of Wilmington, LLC, Wilmington, North Carolina
  - Accellacare Research of Winston Salem, Winston-Salem, North Carolina
  - Diabetes and Endocrinology Associates of Stark County, Inc., Canton, Ohio
  - Tekton Research, Edmond, Oklahoma
  - Roper St. Francis Physician Partners - Primary Care, Mt. Pleasant, South Carolina
  - Norwood Family Medicine, Knoxville, Tennessee
  - Summit-Halls Family Practice, Knoxville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Velocity Clinical Research - Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center Investigation Drug Services, Dallas, Texas
  - Juno Research, LLC, Houston, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Privia Medical Group North Texas - Stephenville, Stephenville, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
- Centro Medico Viamonte SRL, Buenos Aires, Provincia de Buenos, Argentina
- Canada (2):
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Aggarwal and Associates, Brampton, Ontario
- Mexico (9):
  - CEMDEC S.A. de C.V., Cuauhtémoc
  - Instituto de Diabetes Obesidad y Nutricion, SC, Cuernavaca
  - SINACOR, Culiacán
  - Centro De Investigacion En Artritis Y Osteopososis, Mexicali
  - Clinicos Asociados Bocm, S.C., Mexico City
  - Medical Care and Research S.A de C.V, Mérida
  - Avant Santé Research Center, San Pedro Garza García
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
  - FAICIC S de R.L. de C.V, Veracruz
- New Zealand (5):
  - Optimal Clinical Trials - North, Rosedale, Auckland
  - Momentum Pukekohe, Auckland
  - Optimal Clinical Trials, Grafton
  - Tauranga Hospital, Tauranga
  - Momentum Wellington, Wellington
- ISIS Clinical Research Center, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No